CLINICAL TRIAL: NCT00185484
Title: Multi-center, Open, Uncontrolled Study to Investigate the Efficacy and Safety of the Oral Contraceptive SH T 186 D Containing 0.02 mg Ethinylestradiol-b-cyclodextrin Clathrate and 3 mg Drospirenone in a 24-day Regimen for 13 Cycles in 1010 Healthy Female Volunteers
Brief Title: Efficacy and Safety Oral Contraceptive Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91353; 308021
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Contraception
Keywords: Oral contraception
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: YAZ (DRSP 3 mg/EE 0.02 mg, BAY86-5300)

INTERVENTIONS:
Drug: YAZ (DRSP 3 mg/EE 0.02 mg, BAY86-5300) — Oral administration of YAZ (0.02mg ethinyl estradiol-ß-cyclodextrin clathrate and 3mg drospirenone, 24 day hormone tablets followed by 4 days of placebo tablets for 13 cycles

SUMMARY:
The purpose of this study is to determine whether the study drug is effective in prevention of pregnancy in healthy women in reproductive age

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman requesting contraception
* Age between 18 and 35 years (inclusive), smokers maximum age of 30 years (inclusive)

Exclusion Criteria:

* Any conditions might interfere study outcome

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1113 (Actual)
Dates: Start 2004-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Rate of unintended pregnancies (Pearl index) | 13 cycles of 28 days

SECONDARY OUTCOMES:
Physical and gynecological examination | screening, cycle 6 and final examination
Vital signs | each visit
Body weight | each visit
Cervical smear | each visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- [Result] Anttila L, Neunteufel W, Petraglia F, Marr J, Kunz M. Cycle control and bleeding pattern of a 24/4 regimen of drospirenone 3 mg/ethinylestradiol 20 mug compared with a 21/7 regimen of desogestrel 150 mug/ethinylestradiol 20 mug: a pooled analysis. Clin Drug Investig. 2011;31(8):519-525. doi: 10.2165/11590260-000000000-00000. PMID 21721590
- [Result] Anttila L, Bachmann G, Hernadi L, Kunz M, Marr J, Klipping C. Contraceptive efficacy of a combined oral contraceptive containing ethinyloestradiol 20 mug/drospirenone 3mg administered in a 24/4 regimen: a pooled analysis of four open-label studies. Eur J Obstet Gynecol Reprod Biol. 2011 Apr;155(2):180-2. doi: 10.1016/j.ejogrb.2010.12.037. Epub 2011 Feb 1. PMID 21277674